CLINICAL TRIAL: NCT06391190
Title: A Prospective Single Arm Trial of Concurrent Chemoradiotherapy (With Albumin-Bound Paclitaxel/Cisplatin) Followed by PD-1 Inhibitor in Locally Advanced Cervical Cancer
Brief Title: Concurrent Chemoradiotherapy Followed by PD-1 Inhibitor in Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACCI
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Cervical Carcinoma; Concurrent Chemoradiotherapy; Immunotherapy
MeSH Terms: interventions — Albumin-Bound Paclitaxel; Cisplatin; sintilimab; Radiation

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): with Albumin-Bound Paclitaxel 50-75mg/m2, cisplatin 25-40 mg/m2 weekly for up to 5 cycles during radical radiation (EBRT followed by brachytherapy); followed by Sintilimab 200mg Q3W for 8 cycles.
  Interventions: Drug: Albumin-Bound Paclitaxel, cisplatin, Sintilimab

INTERVENTIONS:
Drug: Albumin-Bound Paclitaxel, cisplatin, Sintilimab — with Albumin-Bound Paclitaxel 50-75mg/m2, cisplatin 25-40 mg/m2 weekly for up to 5 cycles during radical radiation; followed by Sintilimab 200mg Q3W for 8 cycles
  Other Names: radiation

SUMMARY:
To explore the safety and efficacy of Albumin-Bound Paclitaxel/Platinum based concurrent chemoradiotherapy Followed by PD-1 inhibitor (Sintilimab) in locally advanced cervical cancer

DETAILED DESCRIPTION:
Patients with pathologically confirmed locally advanced cervical cancer will be treated with concurrent chemoradiotherapy (weekly Albumin-Bound Paclitaxel and cisplatin), followed by Sintilimab 200mg q3w for 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75;
2. Untreated patients with pathologically proven locally advanced cervical cancer;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1
4. Adequate hematological, renal and hepatic functions:

   4.1 Hemoglobin > 8.0 g/dl 4.2 Neutrophils > 2000 cells/μl; Leukocytes > 4 × 109/L 4.3 Platelets > 100 × 109/Lg. 4.4 Serum urea nitrogen (BUN) ≤ 1.5 × upper normal limit (UNL) 4.5 Serum creatinine (Cr) ≤ 1.5 × upper normal limit (UNL) 4.6 Serum ALT/AST ≤ 2.5× UNL 4.7 Serum Total bilirubin ≤ 1.5× UNL
5. Life expectancy > 6 months
6. Eligible for concurrent chemoradiotherapy assessed by principle investigator;
7. No obvious active bleeding;
8. Written informed consent must be available before study registration.

Exclusion Criteria:

1. Recurrent or distant metastatic disease;
2. Prior malignancies (other than curable non-melanoma skin cancer) within 5 years;
3. Active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of substantial amount of hormones or other immunosuppressants;
4. Patients who need to receive systemic corticosteroids (dose equivalent to or higher than prednisone 10mg qd) or other immunosuppressants within 14 days before enrollment or during the study;
5. Vaccination of live attenuated vaccine 30 days before enrollment, or planned vaccination of live attenuated vaccine during the study;
6. Previous organ transplantation or HIV patients;
7. Allergic to macromolecular proteins /monoclonal antibodies, or to any test drug component;
8. Active acute or chronic viral hepatitis B or C. Hepatitis B virus (HBV) DNA> 2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA> 103 copies/ml.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
progression disease free survival | -2 years
  the time interval from the date of treatment to disease progression, local or distant recurrence.
safety of Albumin-Bound Paclitaxel/cisplatin based concurrent chemoradiotherapy followed by Sintilimab | -1 years
  the occurrence and grade of side effect from treatment according to the CTCAE 4.0 and NCCN clinical practice guidelines in the evaluation treatment-related toxicity (through the symptoms, physical examination, and also through blood/image/encoscopy examination, such as blood routine, liver and renal function, TSH/T3/T4/ACTH concentration, myocardial enzymes, and EKG, echocardiography, CT, et al).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 months
  the percentage of the participants in the population who have a Complete Response or Partial Response accordingly to RECIST 1.1
distant-metastasis free survival | -2 years
  the time interval from the date of treatment to distant recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- RenJi hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No